CLINICAL TRIAL: NCT00383162
Title: A Study of Combination Product (Sumatriptan Succinate and Naproxen Sodium) in Migraine Subjects Who Report Poor Response or Intolerance to Short Acting Triptans (Study 1 of 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TRX106571
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Results first posted 2010-02-17 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Migraine Disorders
Keywords: Combination Product; naproxen sodium; sumatriptan succinate; short acting triptan; migraine, acute; Poor response
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Product - Placebo (Other): Combination product (sumatriptan and naproxen sodium) [Attack 1] followed by placebo [Attack 2]
  Interventions: Drug: Combination Product (sumatriptan succinate / naproxen sodium); Drug: Placebo
- Placebo - Combination Product (Other): Placebo [Attack 1] followed by Combination Product (sumatriptan and naproxen sodium) [Attack 2]
  Interventions: Drug: Combination Product (sumatriptan succinate / naproxen sodium); Drug: Placebo

INTERVENTIONS:
Drug: Combination Product (sumatriptan succinate / naproxen sodium) — Bilayer tablet containing 85mg sumatriptan (as 119mg sumatriptan succinate; fast disintegrating/rapid release formulation) active ingredient in one layer, and 500mg naproxen sodium active ingredient in the second layer.
Drug: Placebo — Matching placebo tablet.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, crossover, two-attack, out-patient, early-intervention evaluation of subjects who have migraine with or without aura and who discontinued use of short acting triptan(s) within the past year due to non-response or intolerance. Subjects will treat 2 separate migraine attacks during the mild phase of each attack; one attack will be treated with one tablet of the Combination Product (sumatriptan succinate and naproxen sodium) and the other attack with one tablet of placebo (crossover design). [Study 1 of 2]

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, crossover, two-attack, out-patient, early-intervention evaluation of subjects who have migraine with or without aura and who discontinued use of short acting triptan(s) within the past year due to non-response or intolerance. Subjects will treat 2 separate migraine attacks during the mild phase of each attack; one attack will be treated with one tablet of the Combination Product (sumatriptan succinate and naproxen sodium) and the other attack with one tablet of placebo (crossover design); however, the order of these treatments will be randomized. A minimum 1-week washout period is required between study medication treatment of the first and second migraine attacks.

Each subject will have two visits: (1) a Screening visit at study entry and (2) a Final visit 4-10 days after the second (or last) attack. A telephone contact will also be required 1-3 days after the first attack, and then once per month until the Final visit.

The primary study objective is to assess efficacy as measured by sustained pain-free (SPF) relief of Combination Product compared to placebo in treating migraine subjects who have previously discontinued treatment with short acting triptans (rizatriptan, sumatriptan, almotriptan, zolmitriptan, and eletriptan).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female between 18 and 65 years old.
* Subject has migraine with or without aura (2004 ICHD-II criteria).
* Subject has 1-8 migraines per month over the previous 3 months and less than 15 total headache days per month.
* Subject has recently (within 1 year) discontinued the use of eletriptan, rizatriptan, sumatriptan, almotriptan, or zolmitriptan, due to nonresponse or intolerable adverse events. Non-response is defined as documented discontinuation of treatment with eletriptan, rizatriptan, sumatriptan, almotriptan, or zolmitriptan for reasons related to response, including (but not limited to): slow onset of efficacy, inconsistent efficacy, inadequate overall efficacy, or inadequate sustained efficacy through 24 hours. Intolerance is defined as documented discontinuation of treatment with eletriptan, rizatriptan, sumatriptan, almotriptan, or zolmitriptan for other reasons, attributable to the triptan, outside of non-response.

A female is eligible to enter and participate in this study if she is of:

* non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
* child-bearing potential, has a negative urine pregnancy test at screen, and agrees to one of the following acceptable measures of contraception:
* Complete abstinence from intercourse from 2 weeks prior to administration of the investigational product, throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the investigational drug (a minimum of 5 days); subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit; or,
* Female sterilization; or,
* Sterilization of male partner; or,
* Implants of levonorgestrel; or,
* Injectable progestogen; or,
* Oral contraceptive (combined or progestogen only); or,
* Any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year (not all IUDs meet this criterion); or,
* Spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a female diaphragm); or,
* Any other methods with published data showing that the highest expected failure rate for that method is less than 1% per year; or,
* Any other barrier methods only if used in combination with any of the above acceptable methods.
* Subject taking oral contraceptives has been on a stable regimen for at least 2 months prior to screening.
* Subject is willing and able to provide informed consent prior to entry into this treatment phase of the study.
* Subject is able to understand and complete the diary card.

Exclusion Criteria: Subjects with any of the following criteria may not enroll in the study:

* Subject has non-migraine headache, retinal migraine, basilar or hemiplegic migraine, cluster headache, or headaches secondary to trauma, cranial or cervical disorders, infections, alterations of homeostasis, ENT disorders, psychiatric disorders or cranial neuralgias.
* Subject has confirmed or suspected ischemic heart disease (angina pectoris, history of myocardial infarction, documented silent ischemia), Prinzmetal's angina/coronary vasospasm, or signs/symptoms consistent with any of the above.
* Subject has evidence or history of ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome.
* Subject has cardiac arrhythmias requiring medication or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in this study.
* Subject has a history of cerebrovascular pathology including stroke and/or transient ischemic attacks (TIAs).
* Subject has a history of congenital heart disease.
* Subject has uncontrolled hypertension at screening (sitting systolic pressure ≥140mmHg, diastolic pressure ≥90mmHg).
* Subject, in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease (based on history or the presence of risk factors including but not limited to, hypertension, hypercholesterolemia, smoker, obesity, diabetes, strong family history of coronary artery disease, female with surgical or physiological menopause, or male over 40 years of age).
* Subject has a history of epilepsy or structural brain lesions which lower the convulsive threshold or treated with an antiepileptic drug for seizure control within 5 years prior to screening.
* Subject has a history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study.
* Subject is currently taking a monoamine oxidase inhibitor (MAOI), or has taken a MAOI within 2 weeks prior to screening or plans to take within 2 weeks after treatment.
* Subject is currently taking, or has taken in the previous three months, a migraine prophylactic medication containing methysergide or dihydroergotamine; or is taking a medication that is not stabilized (i.e. change of dose within the past 2 months) for either chronic or intermittent migraine prophylaxis or for a co-morbid condition that is not stabilized..
* Subject is currently taking any anti-coagulant (e.g., warfarin).
* Subject has a recent history of regular use of opioids or barbiturates for treatment of their migraine headache and/or other non-migraine pain. Regular use is defined as an average of 4 days per month over the last 6 months.
* Subject is currently taking or has taken in the previous 4 weeks, herbal preparations containing St. John's Wort (Hypericum perforatum).
* Subject has hypersensitivity, intolerance, or contraindication to the use of sumatriptan or naproxen sodium or any of their components or any other 5-HT1 receptor agonist.
* Subject has a history of allergic reactions to naproxen preparations, including subject in whom aspirin or other NSAID drugs induce the syndrome of asthma, rhinitis, and nasal polyps.
* Subject has a history of any gastrointestinal surgery that specifically indicates a past history of bleeding, ulceration or perforation.
* Subject has a history of gastric bypass or stapling surgery.
* Subject has a history of GI ulceration in the past six months or gastrointestinal bleeding in the past year.
* Subject has a history of inflammatory bowel disease.
* Subject has a history of any bleeding disorder.
* Subject is taking any antiplatelet agent (except low-dose aspirin ≤ 325mg/day for cardioprotective reasons).
* Subject is taking any angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker.
* Subject is pregnant, actively trying to become pregnant or breast-feeding.
* Subject has evidence of alcohol or substance abuse within the last year which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results.
* Subject has any concurrent medical or psychiatric condition which, in the investigator's opinion, may affect the interpretation of efficacy and safety data or which otherwise contraindicates participation in this clinical trial.
* Subject has participated in an investigational drug trial within the previous four weeks or plans to participate in another study at any time during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (26):
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Fairfield, Connecticut
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Northbrook, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Orchard Park, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Matthews, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Mathew N, Landy S, Tietjen G, Stark S, Runken M, Lener S, Derosier F, and Bukenya D. Evaluation of a single fixed-dose tablet of Sumatriptan 85 mg formulated with RT Technology/Naproxen sodium 500 mg (SumaRT/Nap) in Subjects who Reported Poor Response or Intolerance to Short Acting Triptans for the Acute Treatment of Migraine. Headache 2008: S44-45.
- [Background] Mathew NT, Landy S, Stark S, Tietjen GE, Derosier FJ, White J, Lener SE, Bukenya D. Fixed-dose sumatriptan and naproxen in poor responders to triptans with a short half-life. Headache. 2009 Jul;49(7):971-82. doi: 10.1111/j.1526-4610.2009.01458.x. Epub 2009 May 27. PMID 19486178
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: TRX106571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: TRX106571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TRX106571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: TRX106571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TRX106571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TRX106571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TRX106571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Sumatriptan-Naproxen: Participants who were randomized to treat the first of two migraine attacks with Placebo (period 1) and the second attack with 85 mg/Naproxen Sodium 500 mg (period 2).
- Sumatriptan-Naproxen/Placebo: Participants who were randomized to treat the first of two migraine attacks with 85 mg/Naproxen Sodium 500 mg (period 1) and the second attack with Placebo (period 2).
Period: Migraine Attack 1 (Period 1)
Arm/Group | Placebo/Sumatriptan-Naproxen | Sumatriptan-Naproxen/Placebo
Started | 87 | 86
Completed | 67 (Participants completing a period treated a migraine with investigational product.) | 73 (Participants not completing did not take investigational product.)
Not Completed | 20 | 13
Not completed — No opportunity to treat migraine | 3 | 4
Not completed — Lost to Follow-up | 8 | 7
Not completed — Did not meet eligibility criteria | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Non-compliant | 3 | 0
Period: Migraine Attack 2 (Period 2)
Arm/Group | Placebo/Sumatriptan-Naproxen | Sumatriptan-Naproxen/Placebo
Started | 67 | 73
Completed | 65 | 66
Not Completed | 2 | 7
Not completed — No opportunity to treat migraine 2 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Unknown reason | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: Safety Population - Participants who were randomized and who treated at least 1 migraine attack with investigational product.
Arm/Group | Safety Population
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.34)
Gender [Count of Participants; unit: Participants]
  Female | 122
  Male | 22
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian/European heritage | 132
  African American/African Heritage | 5
  East Asian Heritage | 1
  South East Asian Heritage | 2
  Arabic/North African Heritage | 1
  Mixed Race | 1
  Other - Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Sustained Freedom From Migraine Pain Between 2-24 Hours Post-dose
Description: Sustained freedom from migraine pain was defined as having no pain at 2 hours post-dose without the use of rescue medication; and without the recurrence of any pain or the use of any rescue medication 2 to 24 hours post-dose.
Time Frame: 2 - 24 hours post-dose
Population: Intent-to-Treat (ITT) population included subjects in the Safety Population who provided an evaluation of their Investigational Product (IP) for at least one treated attack.
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 10 | 36
Statistical Analysis 1: Comparison: Placebo vs Sumatriptan-Naproxen Sodium; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations; Odds Ratio (OR) = 4.50, 95% CI [2.17 to 9.36]

2. Secondary Outcome: Pain-Free Assessment at 2 Hours Post-dose
Description: Participants rated their pain severity using a four point scale where 0=no pain, 1=mild pain, 2=moderate pain, and 3=severe pain. Pain-free was a rating of 0 (no pain) at the specified time.
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 23 | 54

3. Secondary Outcome: Rescue Medication Used up to 24 Hours Post-dose
Description: A rescue medication was defined as an additional medication taken for the treatment of migraine headache pain symptoms associated with the attack. Allowed were a single dose of either: sumatriptan (50mg or 100mg), OR naproxen sodium (max 550mg), OR, an over-the-counter pain-reliever (per label).
Time Frame: Dosing to 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 84 | 40

4. Secondary Outcome: Pain-Free Assessment at 1/2, 1, 4, 8 Hours Post-dose
Description: as for outcome 2
Time Frame: 1/2, 1, 4, and 8 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants
  1/2 hour post-dose | 2 | 6
  1 hour post-dose | 13 | 26
  4 hours post-dose | 30 | 80
  8 hours post-dose | 32 | 88

5. Secondary Outcome: Sustained Freedom From Migraine
Description: Migraine-free was defined as pain-free with no traditional migraine-associated symptoms (i.e.,photophobia, phonophobia, nausea). Sustained migraine-free was defined as migraine-free at 2 hours and sustained from 2 to 24 hours post dose without the use of rescue medication.
Time Frame: 2 - 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 11 | 32

6. Secondary Outcome: Migraine-Free Assessment at 2, 4, and 8 Hours Post-dose
Description: Migraine-free was defined as pain-free with no traditional migraine-associated symptoms (i.e.,photophobia, phonophobia, nausea and vomiting) at the time of the assessment.
Time Frame: 2, 4 , and 8 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants
  2 hours post-dose | 19 | 47
  4 hours post-dose | 30 | 72
  8 hours post-dose | 29 | 80

7. Secondary Outcome: Sustained Freedom From Migraine-Associated Sinus Pain
Description: Sustained Freedom from Migraine-Associated Sinus Pain was defined as the absence of sinus pain from 2 to 24 hours post-dose.
Time Frame: 2 - 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 34 | 76

8. Secondary Outcome: Migraine-Associated Sinus Pain Assessed at Baseline, 2, 4, and 8 Hours Post-dose
Description: Number of participants who had sinus pain at the time of assessment.
Time Frame: Baseline, 2, 4, and 8 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants
  Baseline | 58 | 61
  2 hours post-dose | 52 | 31
  4 hours post-dose | 39 | 20
  8 hours post-dose | 35 | 19

9. Secondary Outcome: Sustained Freedom From Migraine-Associated Neck Pain
Description: Sustained Freedom from Migraine-Associated Neck Pain was defined as the absence of neck pain from 2 to 24 hours post-dose.
Time Frame: 2 - 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 33 | 63

10. Secondary Outcome: Migraine-Associated Neck Pain Assessed at Baseline, 2, 4, and 8 Hours Post-dose
Description: Number of Participants with neck pain at the time of assessment.
Time Frame: Baseline, 2, 4, and 8 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants
  Baseline | 65 | 82
  2 hours post-dose | 54 | 54
  4 hours post-dose | 46 | 40
  8 hours post-dose | 37 | 31

11. Secondary Outcome: Sustained Freedom From Migraine-Associated Photophobia
Description: Sustained Freedom from Migraine-Associated Photophobia was defined as the absence of photophobia (sensitivity to light) from 2 to 24 hours post-dose.
Time Frame: 2 - 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 23 | 59

12. Secondary Outcome: Migraine-Associated Photophobia Assessed at Baseline, 2, 4, and 8 Hours Post-dose
Description: Number of participants who had photophobia (sensitivity to light) at the time of assessment.
Time Frame: Baseline, 2, 4, and 8 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants
  Baseline | 98 | 95
  2 hours post-dose | 86 | 57
  4 hours post-dose | 65 | 33
  8 hours post-dose | 48 | 27

13. Secondary Outcome: Sustained Freedom From Migraine-Associated Phonophobia
Description: Sustained Freedom from Migraine-Associated Phonophobia was defined as the absence of phonophobia (sensitivity to noise) from 2 to 24 hours post-dose.
Time Frame: 2 - 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 31 | 66

14. Secondary Outcome: Migraine-Associated Phonophobia Assessed at Baseline, 2, 4, and 8 Hours Post-dose
Description: Number of participants who had phonophobia (sensitivity to noise) at the time of assessment.
Time Frame: Baseline, 2, 4, and 8 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants
  Baseline | 82 | 86
  2 hours post-dose | 73 | 47
  4 hours post-dose | 56 | 31
  8 hours post-dose | 44 | 24

15. Secondary Outcome: Sustained Freedom From Migraine-Associated Nausea
Description: Sustained Freedom from Migraine-Associated Nausea was defined as the absence of nausea from 2 to 24 hours post-dose.
Time Frame: 2 - 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 38 | 70

16. Secondary Outcome: Migraine-Associated Nausea Assessed at Baseline, 2, 4, and 8 Hours Post-dose
Description: Number of participants who had nausea at the time of assessment. Resolution of an associated symptom was defined as a migraine headache symptom that was present at the time of treatment that was not present post-dose. Symptom resolution was defined only among subjects who treated while their symptom was present.
Time Frame: Baseline, 2, 4, and 8 hours
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants
  Baseline | 45 | 48
  2 hours post-dose | 42 | 39
  4 hours post-dose | 29 | 20
  8 hours post-dose | 24 | 14

17. Secondary Outcome: Sustained Complete Pain/Symptom-Free
Description: Sustained Complete Pain/Symptom-Free was defined as completely symptom-free (migraine-free plus neck and sinus pain-free) at 2 hours and sustained from 2 to 24 hours without the use of rescue medication.
Time Frame: 2 - 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants | 9 | 30

18. Secondary Outcome: Complete Pain/Symptom-Free Assessed at Baseline, 2, 4, and 8 Hours Post-dose
Description: Number of participants who were completely symptom-free (migraine-free plus neck and sinus pain-free) at time of assessment."Complete pain/symptom-free" was defined as migraine-free, neck pain-free, and sinus pain free.
Time Frame: Baseline, 2, 4, and 8 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 133 | 136
Participants
  Baseline | 133 | 136
  2 hours post-dose | 117 | 92
  4 hours post-dose | 107 | 73
  8 hours post-dose | 106 | 62

19. Secondary Outcome: Recurrence of Any Migraine Headache Pain
Description: Recurrence is defined as the return of any migraine headache pain during the specified post-dose period, following a pain-free response at 2 hours.
Time Frame: 24 hours and 48 hours
Population: Subpopulation of the Intent-to-Treat population of subjects who were pain-free at 2 hours post-dose. Placebo-23 subjects and Sumatriptan/Naproxen Sodium 54 subjects
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Number analyzed (Participants) | 23 | 54
Participants
  Recurrence by 24 hours post-dose | 12 | 11
  Recurrence by 48 hours post-dose | 13 | 11

ADVERSE EVENTS:
Groups:
- Placebo: Subjects who were randomized to take Placebo during Migraine period 1, then a one week wash-out period without any drugs, and then given Sumatriptan 85 mg/Naproxen Sodium 500 mg during Migraine period 2.
- Sumatriptan-Naproxen Sodium: Subjects who were randomized to take Sumatriptan 85 mg/Naproxen Sodium 500 mg during Migraine period 1, then a one week wash-out period without any drugs, and then given Placebo during Migraine period 2.
Arm/Group | Placebo | Sumatriptan-Naproxen Sodium
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/140
Other Adverse Events (participants affected / at risk) | 0/135 | 0/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.